CLINICAL TRIAL: NCT00182247
Title: D-Dimer and IPG for Recurrent Thrombosis (DIRECT) Study
Brief Title: D-Dimer and IPG for Recurrent Thrombosis (DIRECT)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: Heart and Stroke Foundation of Canada (Other)
Organization: McMaster University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CTMG-1998-DIRECT
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2005-09-16 (Estimated); Status verified 2005-09

CONDITIONS: Deep Vein Thrombosis; Pulmonary Embolism
Keywords: deep vein thrombosis; DVT; pulmonary embolism; PE; venous thromboembolism; VTE; d-dimer; IPG
MeSH Terms: conditions — Venous Thrombosis; Pulmonary Embolism; Venous Thromboembolism

INTERVENTIONS:
Procedure: venogram

SUMMARY:
To simplify and improve the diagnostic approach to patients with clinically suspected recurrent DVT by determining whether the results of the combination of IPG and d-dimer testing, using a whole blood agglutination assay, can be used in the management of such patients.

ELIGIBILITY:
Inclusion Criteria:

* suspected deep vein thrombosis
* history of previous DVT or PE

Exclusion Criteria:

* comorbid condition limiting survival to less than 6 months
* contraindication to contrast medium (allergy, renal dysfunction, creatinine > 150mcmol/L)
* receiving long-term warfarin or heparin therapy
* received full-dose heparin therapy for more than 48 hours
* pregnancy
* symptomatic for pulmonary embolism
* absence of symptoms within 5 days of presentation
* geographic inaccessibility which precludes follow-up

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 600
Dates: Start 1998-12; Study Completion 2001-01

PRIMARY OUTCOMES:
symptomatic DVT and PE in follow-up

SECONDARY OUTCOMES:
death
deep vein thrombosis diagnosed by venography in those
randomized to that intervention

CONTACTS AND LOCATIONS:
Overall Officials: Shannon Bates, M.D., Study Chair — Hamilton Health Sciences Corporation; Jeffrey Ginsberg, M.D., Principal Investigator — Hamilton Health Sciences Corporation
Locations (8):
- Canada (7):
  - Hamilton General Hospital, Hamilton, Ontario
  - McMaster University Medical Centre, Hamilton, Ontario
  - St. Joseph' Hospital, Hamilton, Ontario
  - Henderson General Hospital, Hamilton, Ontario
  - Chedoke Hospital, Hamilton, Ontario
  - London Health Sciences Centre, London, Ontario
  - CHA - Pavillon Saint-Sacrement, Québec, Quebec
- IRCCS Policlinico S. Matteo, Pavia, Italy